CLINICAL TRIAL: NCT02145026
Title: A Prospective Open-Label Study of the Effectiveness of Epoetin Beta for Treating Anemic Patients With Low/Intermediate-1-Risk Myelodysplastic Syndrome (MDS)
Brief Title: A Study of Epoetin Beta Treatment in Anemic Participants With Myelodysplastic Syndrome (MDS)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML29005
Record Dates: First submitted 2014-05-20; First posted 2014-05-22 (Estimated); Results first posted 2020-04-24 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Myelodysplastic Syndromes
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — epoetin beta

ARMS (1):
- Epoetin Beta (Experimental): Participants will receive epoetin beta at an initial dose of 30,000 International Units (IU) per week administered subcutaneously (SC). Response will be firstly evaluated at Week 4 and the subsequent dose will be based on the response: if hemoglobin level reaches greater than or equal to (>/=)12 grams per deciliter (g/dL) at any time, epoetin beta will be discontinued until hemoglobin levels are less than or equal to (</=) 10 g/dL; if the hemoglobin level increases less than (<) 1 g/dL from screening level and hemoglobin level ˂12 g/dL, a 60,000 IU per week epoetin beta will be administered SC until Week 12; if the hemoglobin level increases >/=1 g/dL from screening level and hemoglobin level ˂12 g/dL, a 30,000 IU per week epoetin beta will be continued until Week 12.
  Interventions: Drug: Epoetin beta

INTERVENTIONS:
Drug: Epoetin beta — Epoetin beta 30,000 or 60,000 IU per week SC injection
  Other Names: Recormon

SUMMARY:
This is a Phase IV, prospective, multi-center, open-label study to assess the effectiveness and safety profile of epoetin beta (Recormon®) for treatment of symptomatic anemia in adult participants associated with low/intermediate-1-risk MDS. After screening, eligible participants will be treated with epoetin beta as recommended in the approved label and international guidelines for the use of epoetin in MDS participants and the dosage will be adjusted on the basis of erythroid response.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants with low or intermediate-1 risk MDS
* No previous treatment with hematopoietic growth factors within 3 months prior to screening
* Symptomatic anemia (hemoglobin <10 g/dL) as determined by investigator
* Serum erythropoietin <500 milliunits/milliliter (mU/mL) within 14 days prior to the first dose of study treatment
* Require no red blood cell transfusion or dependent on <4 units within 8 weeks prior to screening
* Clinically stable for at least 1 month prior to entry into the study
* For female participants of childbearing potential and male participants with partners of childbearing potential, agreement (by participants and/or partner) to use highly effective form(s) of contraception

Exclusion Criteria:

* Contraindications and/or known hypersensitivity to the active substance and/or any of the excipients of epoetin beta treatment
* Poorly controlled hypertension as assessed by the investigator
* History of Acute Myeloid Leukemia (AML) or high risk for AML
* Administration of another investigational drug within 1 month before screening or planned during the study period
* Previously documented evidence of Pure Red Cell Aplasia (PRCA)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-08-06 (Actual); Primary Completion 2019-04-09 (Actual); Study Completion 2019-04-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (10):
- Thailand (10):
  - King Chulalongkorn Memorial Hospital; Division of Hematology, Department of Medicine, Bangkok
  - Rajavithi Hospital; Medicine, Bangkok
  - Ramathibodi Hospital; Division of Hematology, Department of Medicine, Bangkok
  - Siriraj Hospital; Division of Hematology, Department of Medicine, Bangkok
  - Chiang Mai Uni Hospital; Division of Hematology,Dept of Medicine,Faculty of Medicine, Chiang Mai
  - Khonkean Regional Hospital; Medicine, Khon Kaen
  - Srinagarind Hospital, Khon Kaen Uni ; Dept of Medicine, Khon Kaen
  - Thammasart Chalermprakiert Hospital, Thammasart Uni; Hematology, Pathum Thani
  - Naresaun University hospital, Phitsanulok
  - Sapprasitthiprasong Hospital, Ubon Ratchathani

RESULTS

PARTICIPANT FLOW:
Groups:
- Epoetin Beta: Participants received epoetin beta at an initial dose of 30,000 International Units (IU) per week administered subcutaneously (SC). Initial response was evaluated at Week 4 and the subsequent dose was based on response: for hemoglobin levels >/= 12 grams per deciliter (g/dL), epoetin beta was discontinued until levels were </= 10 g/dL; for hemoglobin levels <12 g/dL and that increased less than 1 g/dL, 60,000 IU of epoetin beta were administered until Week 12; and for hemoglobin levels <12 g/dL and that increased >/= 1 g/dL, 30,000 IU of epoetin beta were administered until Week 12.
Period: Overall Study
Arm/Group | Epoetin Beta
Started | 100
Completed | 88
Not Completed | 12
Not completed — Adverse Event | 2
Not completed — Death | 4
Not completed — Withdrawal by Subject | 2
Not completed — Physician Decision | 4

BASELINE CHARACTERISTICS:
Population: 1 participant withdrew at the baseline visit prior to study treatment and was not included in baseline, safety, and intent-to-treat (ITT) analyses.
Arm/Group | Epoetin Beta
Number analyzed (Participants) | 99
Age, Continuous [Mean (Standard Deviation); unit: Years] | 72.9 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69
  Male | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 99
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 99

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants Achieving Erythroid Response at Week 12 as Assessed by International Working Group (IWG) 2006 Response Criteria
Description: Erythroid response at Week 12 according to IWG 2006 criteria was defined as a hemoglobin (Hb) increase of >/= 1.5 grams/deciliter (g/dL), and a reduction of units of red blood cell (RBC) transfusions by at least 4 transfusions/8 weeks compared with the pre-treatment transfusion number in the previous 8 weeks. Only RBC transfusions given for an Hb of </= 9.0 g/dL pre-treatment were counted in the RBC transfusion response evaluation.
Time Frame: Week 12
Population: Efficacy analysis was performed on the intent-to-treat (ITT) population, defined as all enrolled participants who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Epoetin Beta
Number analyzed (Participants) | 99
Participants | 60

2. Secondary Outcome: Percentage of Participants With Platelet Response (in Participants With Pre-Treatment Platelets <100*10^9 Per Liter) at Week 12 as Assessed by IWG 2006 Response Criteria
Description: Platelet response according to IWG 2006 criteria was defined as an absolute increase of >/= 30x10^9/L for participants starting with >20x10^9/L platelets.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Epoetin Beta
Number analyzed (Participants) | 99
Percentage of Participants | 16

3. Secondary Outcome: Percentage of Participants With Neutrophil Response (in Participants With Pre-Treatment Neutrophil <1.0*10^9 Per Liter) at Week 12 as Assessed by IWG 2006 Response Criteria
Description: Neutrophil response according to IWG 2006 criteria was defined as at least 100% increase and an absolute increase of >0.5x10^9/L.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Epoetin Beta
Number analyzed (Participants) | 99
Percentage of Participants | 33.3

4. Secondary Outcome: Percentage of Participants With Adverse Events
Time Frame: From signing of informed consent up to 4 weeks after last dose (up to 18 weeks)
Population: The safety population included all participants that received at least one dose of study medication.
Measure: Number; unit: Percentage of Participants
Arm/Group | Epoetin Beta
Number analyzed (Participants) | 99
Percentage of Participants | 48.48

ADVERSE EVENTS:
Time Frame: Approximately 56 months
Arm/Group | Epoetin Beta
All-Cause Mortality (participants affected / at risk) | 4/99
Serious Adverse Events (participants affected / at risk) | 21/99
Other Adverse Events (participants affected / at risk) | 48/99
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Epoetin Beta (N=99)
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 1 (2)
Congestive heart failure (Cardiac disorders) | 1 (1)
Cardiac tamponade (Cardiac disorders) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 1 (1)
Tachyarrhythmia (Cardiac disorders) | 1 (1)
Gastrointestinal bleeding (Gastrointestinal disorders) | 1 (1)
Esophageal varices (Gastrointestinal disorders) | 1 (1)
Abscess oral (Infections and infestations) | 1 (1)
Hospital acquired pneumonia (Infections and infestations) | 1 (1)
Lobar pneumonia (Infections and infestations) | 1 (1)
Necrotizing fasciitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Septic shock (Infections and infestations) | 1 (1)
Syphilis (Infections and infestations) | 1 (1)
Recurrent urinary tract infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (2)
Urosepsis (Infections and infestations) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (2)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Hypertension worsened (Vascular disorders) | 1 (1)
Hypertensive emergency (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Epoetin Beta (N=99)
Acute diarrhea (Gastrointestinal disorders) | 1 (1)
Aphthous ulcer (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Short-bowel syndrome (Gastrointestinal disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Eosinophilia (Blood and lymphatic system disorders) | 1 (1)
Anemia aggravated (Blood and lymphatic system disorders) | 1 (1)
Anxiety (General disorders) | 1 (1)
Leg pain (General disorders) | 1 (1)
Lymphatic obstruction (General disorders) | 1 (1)
Closed fracture (General disorders) | 1 (1)
Elevated blood pressure (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Gallstones (General disorders) | 1 (1)
Headache (General disorders) | 1 (1)
Increased blood pressure (General disorders) | 1 (1)
Uric acid level increased (General disorders) | 1 (1)
Insomnia (General disorders) | 3 (3)
Leg edema (General disorders) | 1 (1)
Low back pain (General disorders) | 1 (1)
Epistaxis (General disorders) | 1 (1)
Rash (General disorders) | 1 (1)
Purpura senile (General disorders) | 1 (1)
Vertigo (General disorders) | 1 (1)
Chronic kidney disease (General disorders) | 1 (1)
Chronic gingivitis (Infections and infestations) | 1 (1)
Ecthyma gangrenosum (Infections and infestations) | 1 (1)
Hepres zoster (Infections and infestations) | 1 (1)
Conjunctivitis (Infections and infestations) | 1 (1)
Otitis media (Infections and infestations) | 1 (1)
Rhinitis (Infections and infestations) | 1 (1)
Tinea corporis (Infections and infestations) | 1 (1)
Tinea infection (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 3 (3)
Urinary tract infection (Infections and infestations) | 2 (2)
Alkaline phosphatase increased (Investigations) | 1 (1)
Systolic ejection murmur (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypertension (Vascular disorders) | 6 (6)
Hypertension worsened (Vascular disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
Data for the secondary efficacy endpoints (% of participants with platelet response and % of participants with neutrophil response) is not conclusive given the small number of participants meeting the evaluation criteria for each endpoint.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2016-09-12): https://cdn.clinicaltrials.gov/large-docs/26/NCT02145026/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-21): https://cdn.clinicaltrials.gov/large-docs/26/NCT02145026/SAP_001.pdf